CLINICAL TRIAL: NCT02126917
Title: Single-center, Open-Label, 3-Period Crossover, Phase 1 Study to Evaluate the Pharmacokinetics of Hydrocodone Bitartrate Extended-Release (HC-ER) Capsules 50 mg When Co-Administered With Alcohol in Healthy Subjects Under Fasted Conditions
Brief Title: A Study to Determine the Influence of Co-ingestion of Alcohol on Hydrocodone Bitartrate Extended Release (HC-ER)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZX002-0901
Record Dates: First submitted 2014-04-15; First posted 2014-04-30 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Phase 1; Alcohol; Hydrocodone Bitartrate; Pharmacokinetics
MeSH Terms: interventions — Ethanol; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HC-ER + 40% Alcohol (Experimental): Open-label, single-dose, 3-period cross-over. All patients fulfilling inclusion/exclusion received HC-ER 50 mg capsule with 40% Alcohol.
  Interventions: Drug: HC-ER + 40% Alcohol
- HC-ER + 20% Alcohol (Experimental): Open-label, single-dose, 3-period cross-over. All patients fulfilling inclusion/exclusion received HC-ER 50 mg capsule with 20% Alcohol.
  Interventions: Drug: HC-ER + 20% Alcohol
- HC-ER + 0% Alcohol (Experimental): Open-label, single-dose, 3-period cross-over. All patients fulfilling inclusion/exclusion received HC-ER 50 mg capsule with 0% Alcohol.
  Interventions: Drug: HC-ER + 0% Alcohol

INTERVENTIONS:
Drug: HC-ER + 40% Alcohol — HC-ER 50 mg + 240 mL solution of 40% alcohol/orange juice in fasted state
  Other Names: Zohydro ER
  Arms: HC-ER + 40% Alcohol
Drug: HC-ER + 20% Alcohol — HC-ER 50 mg + 240 mL solution of 20% alcohol/orange juice in fasted state
  Other Names: Zohydro ER
  Arms: HC-ER + 20% Alcohol
Drug: HC-ER + 0% Alcohol — HC-ER 50 mg + 240 mL solution of 0% alcohol/orange juice in fasted state
  Other Names: Zohydro ER
  Arms: HC-ER + 0% Alcohol

SUMMARY:
To determine the influence of co-ingestion of alcohol on HC-ER.

DETAILED DESCRIPTION:
Determine the influence of co-ingestion of alcohol on the safety, pharmacokinetics, and relative bioavailability of HC-ER 50 mg under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 21 to 45.
* Female, must be of non-childbearing potential.
* Non-smokers for at least 3 months or light smokers (less than 10 pack-years).
* History of moderate consumption of between 7-21 units of alcohol per week.
* Weighed at least 65 kg with a BMI ≥19 and ≤35 kg/m2.
* Were medically healthy with no clinically significant abnormalities.
* Voluntarily consented to participate in the study.
* Were prepared to be compliant with the study procedures.

Exclusion Criteria:

* Women who were pregnant or breastfeeding.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* History or presence of alcoholism or drug abuse.
* Hypersensitivity or idiosyncratic reaction to morphine, hydrocodone (Vicodin) or other opioids; naltrexone, naloxone, or other opioid antagonist.
* History of no alcohol intake (alcohol-naive) or less than moderate alcohol intake.
* History of alcohol intake exceeding the equivalence of 21 units/week or exceeding the average of 3 drinks per day.
* Surgery of the gastrointestinal tract which would interfere with absorption of the study drug.
* Taken hepatic enzyme inducing drugs (e.g., Nizoral, Tagamet) within the previous 3 months.
* Taken prescription medications within the previous 14 days or over the counter (OTC) medications within the previous 7 days prior to Day 1 Period 1.
* Sitting blood pressure was less than 110/45 mmHg at screening.
* On a special diet (except for vegetarians who agree to abide by study diet) during the 28 days prior to the first dose and throughout the study.
* Significant blood donation or loss within 56 days prior to first dose of HC-ER.
* Plasma donation within 7 days prior to first dose of HC-ER.
* Hemoglobin value less than 12.0 g/dL.
* Participated in another clinical trial within 28 days prior to first dose of HC-ER.
* Positive urine test for drugs of abuse.
* Positive test for, or had been treated for hepatitis B, hepatitis C or HIV.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Assess the rate and extent of absorption of HC-ER 50 mg capsule following co-ingestion of alcohol under fasted conditions. | Day 1 through Day 18

CONTACTS AND LOCATIONS:
Overall Officials: James Kissling, MD, Principal Investigator — Zogenix, Inc.